CLINICAL TRIAL: NCT06150898
Title: Unravelling the Local and Systemic Effects of Primary Surgery and Perioperative Use of Ketorolac and Pregabalin in Primary Breast Cancer Patients According to Adiposity
Brief Title: Ketorolac and Pregabalin Effects on breaSt Cancer (KePreSt)
Acronym: KePreSt
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IJB-KEPREST-2022
Record Dates: First submitted 2022-03-30; First posted 2023-11-29 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-02

CONDITIONS: Early-stage Breast Cancer; Estrogen-receptor-positive Breast Cancer
Keywords: Surgery; Inflammation; Breast cancer; Neuronal features; Ketorolac; Pregabalin; Adiposity; Neurotransmitter; Nerves
MeSH Terms: conditions — Breast Neoplasms; Inflammation; Obesity | interventions — Specimen Handling; Ketorolac; Tablets; Pregabalin; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- No pre-operative treatment (Experimental): Control group: Standard of care
  Number of subjects: 28 (14 lean patients, defined as Body mass index <25 kg/m², and 14 overweight/obese patients, defined as BMI ≥25 kg/m² )
  Interventions: Procedure: Prospective data and sample collection; Drug: Omeprazole 20mg Capsule
- Pre-operative ketorolac (Experimental): Investigational Medicinal Product (IMP): Ketorolac
  Number of subjects: 28 (14 lean patients, defined as Body mass index <25 kg/m², and 14 overweight/obese patients, defined as BMI ≥25 kg/m² )
  Interventions: Procedure: Prospective data and sample collection; Drug: Ketorolac 10 Mg Oral Tablet; Drug: Omeprazole 20mg Capsule
- Pre-operative pregabalin (Experimental): Investigational Medicinal Product (IMP): Pregabalin
  Number of subjects: 28 (14 lean patients, defined as Body mass index <25 kg/m², and 14 overweight/obese patients, defined as BMI ≥25 kg/m² )
  Interventions: Procedure: Prospective data and sample collection; Drug: Pregabalin 75mg; Drug: Omeprazole 20mg Capsule
- Pre-operative ketorolac and pregabalin (Experimental): Investigational Medicinal Products (IMPs): Ketorolac and pregabalin
  Number of subjects: 28 (14 lean patients, defined as Body mass index <25 kg/m², and 14 overweight/obese patients, defined as BMI ≥25 kg/m² )
  Interventions: Procedure: Prospective data and sample collection; Drug: Ketorolac 10 Mg Oral Tablet; Drug: Pregabalin 75mg; Drug: Omeprazole 20mg Capsule

INTERVENTIONS:
Procedure: Prospective data and sample collection — Core-needle biopsy of the breast (pre-treatment), surgical sample collection (post-treatment), extra collection of blood samples (pre- and post-treatment), measurements of adiposity, lifestyle questionaire
Drug: Ketorolac 10 Mg Oral Tablet — Patients will receive 10 mg film-coated tablets of ketorolac tromethamine three times a day, for five days before the surgery
  Arms: Pre-operative ketorolac; Pre-operative ketorolac and pregabalin
Drug: Pregabalin 75mg — Patients will receive 75 mg of pregabalin hard capsule twice a day, for seven days before the surgery
  Arms: Pre-operative ketorolac and pregabalin; Pre-operative pregabalin
Drug: Omeprazole 20mg Capsule — Patients will receive 20 mg of omeprazole once a day on an empty stomach, for five days before the surgery
  Other Names: Auxiliary medicinal product

SUMMARY:
Out of all proportion to its short duration, the perioperative period is critical in determining the long-term outcome of cancer.

To contribute to a better understanding of the neural and inflammatory mechanisms underlying this issue, we aim to implement a novel intervention based on the preoperative use of non-steroidal anti-inflammatory drugs (NSAIDs) with or without an anti-epileptic drug.

Our goal is to understand and transform the perioperative window from being a facilitator of metastatic progression to arresting and/or eliminating residual disease using repurposing drugs

DETAILED DESCRIPTION:
The perioperative period presents a unique window of therapeutic opportunities to counteract minimal residual growth and dormancy escape of cancer cells. The main physiological disturbances induced by the surgery, that enhance the tumoral growth in the perioperative period, are due to the neuronal and inflammatory signaling.

We propose a therapeutic modelling of the inflammatory and neurological pathways in a phase II trial using ketorolac and pregabalin, alone or in combination. Ketorolac, a non-selective NSAIDs will target cyclooxygenase (COX)-enzymes, while pregabalin, an anti-epileptic drug will regulates the release of neurotransmitters. Moreover, both drugs have an effect on the postoperative pain and pregabalin has anxiolytic property. Thanks to this study, and through specific blockade, we want to understand how nervous and inflammatory systems remodel the tumour and systemic characteristics. To ensure an integrative analysis of those factors, patient's adiposity as well as other confounding variable will be taken into account.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria in order to be eligible for this study:

1. Age ≥ 18 years and ≤ 70 years old
2. Female
3. Weight ≥ 35 kg
4. Histological diagnosis of invasive breast adenocarcinoma that is estrogen receptor positive as per the updated American Society of Clinical Oncology (ASCO) - College of American Pathologists (CAP) guidelines according to local testing with ER-positive is defined as having an immunohistochemistry (IHC) of 1% or more and/or Allred score of 3 or more
5. Tumour size ≥ 1.5 cm, determined by diagnostic ultrasound or MRI/CT scan.
6. Stage I, II or III disease (non-metastatic)
7. In case of multifocal, multicentric unilateral or bilateral breast: Adenocarcinoma tumours are allowed provided that all foci are ER+ according to local testing
8. Subject scheduled for a primary breast cancer surgery
9. Subject is willing to provide plasma/blood and tumour samples for translational research.
10. Subject is willing to provide tissue from a newly obtained core or excisional biopsy of the tumour that should be evaluable for central histological characterization and future molecular testing
11. Subject is willing to take omeprazole and has no contraindication to omeprazole.
12. Have an HEMSTOP score<2 and conventional coagulation screening test within normal limits such as activated partial thromboplastin time (21.6< aPTT >28.7), international normalised ratio (1.31<INR) and platelet count (>100.10³/ml)
13. Women of childbearing potential must agree to use of one highly effective method of contraception prior study entry, during the course of the study and at least one months after the last administration of study treatment.
14. Negative serum pregnancy test for women of childbearing potential (within 30 days before start of treatment)
15. Subject is willing and able to provide written informed consent for the trial

Exclusion Criteria:

Subjects meeting one of the following criteria are not eligible for this study:

1. Subject planned for intraoperative radiotherapy
2. Subject planned for immediate reconstruction
3. Neoadjuvant BC therapy
4. Allergy to any NSAID or gabapentinoïd
5. Known hypersensitivity reactions to the investigational treatments, or any excipients or auxiliary medicinal products or concomitant medications. Hypersensitive to peanut or soya (related to propofol contraindications)
6. Current use of the antidiabetic agent thiazolidinedione (related to interaction with pregabalin), lithium salts, probenecid, pentoxifylline or intensive diuretic therapy.
7. Current NSAID (> twice a week the year prior to diagnosis) or pregabalin use
8. Previous malignant pathology within 5 years prior to inclusion or currently undergoing maintenance therapy. Exceptions include basal cell carcinoma or squamous cell carcinoma of the skin that have undergone potentially curative therapy or in situ cervical cancer.
9. Active or history of peptic ulcer disease or gastro-intestinal bleeding or perforation
10. Pregnancy or lactating women
11. Chronic inflammatory disease as rheumatoid arthritis, uncontrolled asthma, chronic heart failure, chronic obstructive pulmonary disease, cystic fibrosis, inflammatory myopathies (e.g., idiopathic polymyositis, dermatomyositis, inclusion body myositis), inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis), McArdle's disease, multiple sclerosis, lupus, chronic inflammatory demyelinating polyneuropathy, psoriasis, autoimmune thyroiditis as Graves' disease or Hashimoto's thyroiditis (unless previous surgical ablation), myasthenia gravis, vasculitis.
12. Complete or partial nasal polyposis syndrome, Quincke's oedema, bronchospasm, asthma
13. Known chronic infectious disease as active hepatitis B (defined as positive serology for Ac anti-HBc and IgM anti HBc OR Ac anti HBc and Ag HBs), active hepatitis C (defined as positive serology for anti-VHC and positive PCR-VHC) or active tuberculosis (included under treatment)
14. Uncontrolled HIV infection (defined as detectable viral loads by standard clinical assays) or controlled HIV infection (defined undetectable HIV viral loads by standard clinical assays) treated by one of following drugs: Nelfinavir, Atazanavir or Saquinavir (related to interaction with omeprazole).
15. Infection currently treated with one of the following drugs: posaconazole, voriconazole, ketoconazole and rifampicin, unless discontinuation of treatment is planned at least 10 days prior to the start of study treatment AND with complete resolution according to expert opinion (related to interaction with omeprazole)
16. Inadequate liver function (defined as total serum bilirubin ≥ 2 x upper limit of normal (ULN<1.2 mg/dl) - unless documented Gilbert syndrome- AND Alanine Aminotransferase (ALT) ≥ 2 x ULN (ULN <32 UI/l and ULN <33 UI/l, respectively) AND Alkaline phosphatase (ALP) ≥ 2.5 x ULN (ULN=104 UI/l))
17. Cirrhosis or severe hepatitis.
18. Renal impairment (defined as GFR<90ml/min/1.73m² or serum creatinine > 442 μmol/l or > 5 mg/dL) or single kidney or previous renal surgery
19. Subject with history of (severe) renal toxicity with an NSAID
20. Subject with a recent history of operations associated with a high risk of bleeding
21. Previous, ongoing or suspected cardiovascular disease defined as history of ischemic heart disease or heart failure or uncontrolled high blood pressure (Systolic ≥160mmHg and/or diastolic ≥100mmHg) or peripheral arterial disease or cerebrovascular disease
22. Subject with a recent history of surgery associated with a high risk of bleeding
23. Hemostasis disorder as haemophilia, Von Willebrand disease, constitutional thrombopathies or thrombocytopenia (defined as platelet count < 100 000/mm³), current /planned anticoagulant or anti-platelet therapy.
24. Inadequate bone marrow function (defined as absolute neutrophil count <1000/μL and platelet count <100'000/μL)
25. Systemic immunosuppressive treatment (defined as systemic corticotherapy or anti-rejection treatment or interferon therapy) within the 2-years prior diagnosis
26. Psychiatric disease or antipsychotic/ antidepressant use
27. Epilepsy or any current anti-epileptic drug use
28. Obstructive sleep apnea
29. ASA≥3

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2027-04-20 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
To detect a reduced increase in systemic inflammation (from baseline to up to 24 hours after surgery) using peri-operative ketorolac | Up to 24 hours after surgery
  Plasma multiplex technology using cytometric bead arrays
To detect a reduced increase in systemic neurotransmitters (from baseline to up to 24 hours after surgery) using peri-operative pregabalin | Up to 24 hours after surgery
  Liquid Chromatography coupled to tandem Mass Spectrometry (LC-MS/MS)
Change in biomarkers of metastasis at surgery from baseline | At surgery
  Transcriptome profile and bioinformatic analysis
Change in tumoral immune cells recruitment at surgery from baseline | At surgery
  Characterization of Tumour-infiltrating leukocyte subpopulations using RNA sequencing analysis from fresh frozen tissue sections
Change in tumoral neurogenesis at surgery from baseline | At surgery
  Level of neurogenesis markers using RNA sequencing analysis from fresh frozen tissue section
Change in tumoral neurotransmitters level at surgery from baseline | At surgery
  Using RNA sequencing analysis from fresh frozen tissue sections
Change in Peripheral Blood Mononuclear Cells at surgery from baseline | At surgery
  Fluorescence activated cell sorting (FACS) analysis
Change in systemic neuro-inflammatory mediators at surgery from baseline | At surgery
  Plasma multiplex technology using cytometric bead arrays
Change in systemic neurotransmitters at surgery from baseline | At surgery
  Plasma multiplex technology using cytometric bead arrays

SECONDARY OUTCOMES:
Change in anxiety level at surgery from baseline | At surgery
  Generalized Anxiety Disorder - 7 (GAD - 7) Anxiety score (natural number, range[0 - 21]. A score comprised between 0 - 4 indicates a minimal anxiety, 5-9 a mild anxiety, 10-14 a moderate anxiety and a 15-21 in a severe anxiety.
Post-operative pain | Up to 48 hours after surgery
  Consumption of morphine delivered by a programmable patient-controlled analgesia (PCA) infusion pump (number of requested and effectively delivered bolus/ 24h)

OTHER OUTCOMES:
Body Mass Index | The day before surgery
  Calculated: body mass (kg) divided by height squared (m²)
Body composition | The day before surgery
  Calculated from multiple frequency bio-impedance measurements (in %, range [0 - 100])
Waist-to-hip ratio | The day before surgery
  Waist circumference (cm) divided by hip circumference (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Desmedt, PhD, Study Chair — KU Leuven; Imane Bachir, MD, Study Chair — Jules Bordet Institute
Locations (1):
- Institut Jules Bordet, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No